CLINICAL TRIAL: NCT02328872
Title: Compass - Randomized Controlled Trial of 5-yearly Cervical Screening With Primary HPV Testing Versus Cervical Screening With 2.5-yearly Liquid Based Cytology Testing, in HPV-Unvaccinated and HPV-Vaccinated Women in Australia
Brief Title: Compass - Randomised Controlled Trial of Primary HPV Testing for Cervical Screening in Australia
Acronym: Compass
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VCS Foundation (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Marion Saville, Professor, VCS Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Exec-PP-12
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cancer of the Cervix; Cervical Intraepithelial Neoplasia
Keywords: screening; cervical screening; Human Papillomavirus (HPV); cancer prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (HPV Arm) (Experimental): Molecular testing for HPV with partial genotyping for types 16/18, with referral of the HPV16/18-positive group for diagnostic evaluation, and secondary randomisation of women testing positive for other oncogenic HPV infection (not 16/18), to either image-read cytology screening or dual-stained (DS) cytology testing with p16/Ki67 - the "HPV arm". Screening performed 5 yearly.
  Interventions: Device: Molecular testing for HPV
- Control (LBC Arm) (Active Comparator): Image-read liquid based cytology (LBC) screening with reflex HPV triage testing for low grade smears, the "LBC arm." Screening performed 2.5 yearly.
  Interventions: Device: Liquid Based Cytology

INTERVENTIONS:
Device: Molecular testing for HPV — Molecular testing for HPV with a test allowing partial genotyping for separate identification of types 16/18 from cervical samples. The technology used in this trial will be approved by the Therapeutic Goods Administration (TGA) Australia. It will identify the major HPV oncogenic genotypes in a pool and separately identify HPV 16 and 18. It will also satisfy performance criteria for relative sensitivity and specificity compared to Hybrid Capture 2 (HC2 ) as articulated by Meijer et al, 2009, Guidelines for human papillomavirus DNA test requirements for primary cervical cancer screening in women 30 years and older.
  Arms: Intervention (HPV Arm)
Device: Liquid Based Cytology — The liquid based cytology (LBC) used in this trial will be will be approved by the Therapeutic Goods Administration (TGA) Australia for LBC and appropriately validated and (TGA approved) to perform human papillomavirus testing from a cytology sample.
  Arms: Control (LBC Arm)

SUMMARY:
Compass is a randomised controlled trial of primary HPV testing for cervical cancer screening in Australia. A pilot study involving 5,000 women was carried out in 2013-2014. The trial will involve recruiting 76,300 women from primary health clinics. Women aged 25-69, attending for cervical screening or for routine follow-up will be invited to participate in the 2-arm trial. A liquid-based cytology (LBC) sample will be taken from consenting women and sent to VCS Pathology. Women will be randomised in a 1:2 parallel group allocation to LBC and HPV arms using randomisation with the minimisation procedure, with stratification by birth cohort according to whether offered HPV vaccination in Australia's national publicly-funded HPV vaccination program (date of birth >=July 1st 1980 and <1st July 1980). In the LBC (active control) arm, women will undergo 2.5 yearly image read cytology screening with reflex HPV triage testing for low grade cytology. In the HPV (intervention) arm women will undergo 5 yearly HPV screening with partial genotyping enabling separate identification of HPV16 and HPV18 and referral of this group for diagnostic evaluation, and secondary randomisation of "intermediate risk" women testing positive for oncogenic HPV (but not HPV 16 or 18) to either image read LBC screening or dual-stained (DS) cytology testing with p16/Ki67. The laboratory reports issued to practitioners will specify the recommended management for women, according to study arm and test results.Participating women will be flagged and clinical outcomes will be tracked via the Compass Register. Data linkage between the Compass Register and HPV vaccination records held on the Australian Immunisation Register will be performed in order to integrate vaccination and screening histories for trial participants. Participants will be actively followed for an anticipated 5 years from the time of recruitment and the primary outcome is based on the total cumulative detection of CIN3+ after exit testing at 5 years. The anticipated study completion date of March 2027 takes into consideration the final migration of participants to the National Cancer Screening Register and allows for two years to follow-up any intermediate risk results occurring in the last of the recruited trial participants.

DETAILED DESCRIPTION:
Compass is a randomised controlled trial of primary HPV testing for cervical cancer screening versus cytology screening in Australia. A pilot study involving 5,000 women was carried out in 2013-2014. The main trial will involve recruiting 76,300 women from primary health clinics. Women aged 25-69, attending for cervical screening or for routine follow-up will be invited to participate in the 2-arm trial. A liquid-based cytology (LBC) sample will be taken from consenting women and sent to VCS Pathology, at VCS Foundation. On receipt of a woman's first Compass sample at VCS Pathology she will be randomised in a 1:2 parallel group allocation to LBC and HPV arms using randomisation with the minimisation procedure, with stratification by birth cohort according to whether offered HPV vaccination in Australia's national publicly-funded HPV vaccination program (date of birth >=July 1st 1980 and DOB <1st July 1980).

The screening and management algorithms for the two study arms will be as follows:

LBC Arm: 2.5 yearly image-read cytology screening with reflex HPV triage testing for low grade cytology.

HPV Arm: 5 yearly HPV screening for potentially oncogenic types with partial genotyping enabling separate identification of HPV16 and HPV18 and referral of this group for diagnostic evaluation, and secondary randomisation of "intermediate risk" women testing positive for oncogenic HPV (but not HPV 16 or 18) to either image read LBC screening or dual-stained (DS) cytology testing with p16/Ki67.

The laboratory reports issued to practitioners will specify the recommended management for women, according to study arm and test results.

Participating women will be flagged on the Compass Register and invitation letters will be issued 3 months prior to the designated time for re-screening or follow-up. Clinical outcomes (screening test, colposcopy and histology results) will be tracked via the Compass Register. Data linkage between the Compass Register and HPV vaccination records held on the Australian Immunisation Register will be performed in order to integrate vaccination and screening histories for trial participants. Participants will be followed for an anticipated 5 years from the time of recruitment.

Previous trials in unvaccinated populations have demonstrated increased detection of CIN2+ in HPV-screened (or co-tested) women vs. cytology-alone screened women in the baseline screening round, followed by decreased rates of incident CIN3+ in HPV-screened vs. Pap screened women thereafter. This potentially reflects (i) the increased detection of disease at the CIN2 (treatment) threshold at baseline in HPV-screened women, leading to increased prevention of future CIN3 in the group of women treated for CIN2 at baseline; and (ii) the association, demonstrated in multiple cohort studies, between HPV positivity (especially for types 16/18) and the development of CIN3+ in the future. In the Compass trial, HPV-positive women without verified disease at baseline undergo increased surveillance until testing HPV negative.

A total of 36,300 women in the birth cohorts not offered vaccination and 40,000 women in the cohorts offered vaccination, who are presenting for routine screening, will be recruited, to bring the total number recruited to 76,300 (updated August 2019) (with the additional women representing those presenting for routine follow-up and those recruited for a safety monitoring sample). The sample size requirements for the trial are based on assessment of the cumulative proportion of CIN3+ (including CIN3 and invasive cervical cancer) in women who were screen-negative at baseline. A major impact of this study will be value of extended screening intervals in patients who are screen-negative at baseline. Logistically, it would be difficult to randomise patients after baseline screening and as such, the cumulative 5-year CIN3+ rates in baseline screen-negative patients may no longer be strictly comparative. However, this is a critical scientific question and so the trial is powered for this secondary outcome: the cumulative proportion of CIN3+ (including CIN3 and invasive cervical cancer) in screen-negative women, adjusted for censoring after CIN2+ treatment.

The primary outcome is based on the total cumulative detection of CIN3+. Because the primary outcome includes precancer, there remains a potential benefit from early detection in the baseline screening round, and although this benefit is not explicitly factored into the primary outcome it will be highlighted in the assessment of outcomes in baseline screen-negative women (i.e. in the analysis for Secondary Outcome 1). When assessing total cumulative rates of CIN3+, including both the baseline round and longitudinal follow-up in each arm, the follow-up duration is a critical determinant of the expected relative outcomes for CIN3+ when the two arms are compared. A second critical determinant is the disease ascertainment process at trial exit, and a consistent process using a sensitive screening test followed by equivalent referral and management processes must be performed in both arms. Therefore all women enrolled in Compass will be offered HPV exit testing at 5 years (as the standard recommendation for cervical screening in Australia from December 2017, the HPV exit test will also act as a routine cervical screening test).

A Scientific Advisory Committee will advise the investigator team on issues related to protocol, operations and any other issues brought by the investigators to the Committee. An Independent Data Safety and Monitoring Committee (IDSMC) has been configured to monitor the safety of participants in the trial.

Compass is sponsored by the VCS Foundation, a government-funded health promotion charity. The VCS have received equipment and a funding contribution for the Compass trial from Roche Molecular Systems and Ventana Inc USA.

The following technologies have been selected for use in the trial. All devices used in the trial will be listed on the Australian Register of Therapeutic Goods (ARTG) and will be used within their listed approved use. However, during the course of the trial, alternative products may potentially be used, as appropriate, if they fulfil these criteria and if they are successfully pre-qualified at the VCS in accordance with NATA laboratory requirements, and if they satisfy the Quality Assurance Processes currently being established for new technologies to be used in the Renewal National Cervical Screening Program (since alternate ARTG-listed LBC medium and HPV test technologies are available).

Specimen Collection Technology: Samples in the trial will be collected using a liquid-based sample medium. The technology to be used will be PreserveCyt/ThinPrep (Hologic Inc, Bedford MA) (included on the ARTG).

Image read LBC technology: The Hologic Thinprep Imaging (TPI) System will be used for image read analysis (included on the ARTG).

HPV DNA testing technology: Primary HPV DNA testing will be performed using the COBAS 4800 HPV Test (Roche Molecular Systems Inc., Pleasanton, CA (listed on the ARTG) and incorporating:

* Cobas 4800 System, Sample Preparation Kit: c4800 SMPL PREP
* Cobas 4800 System, Amplification/Detection Kit: c4800 HPV AMP/DET
* Cobas 4800 System, Preparation Kit: c4800 LIQ CYT
* Cobas 4800 System, Wash Buffer Kit: c4800 WB

Dual-stained cytology (DS). Analysis of dual stained cytology for p16/Ki-67 markers in the trial will involve use of the CINtec® PLUS kit (VENTANA MEDICAL SYSTEMS, INC., AZ) (this in-vitro diagnostic medical device is included on the ARTG).

ELIGIBILITY:
Inclusion Criteria:

* Australian residents with a cervix, aged 25-69 years who are attending for routine cervical screening. (Note: since April 2016 recruitment has been confined to the younger strata, i.e. women age-eligible for HPV vaccination aged at least 25 and born on or after 1st July 1980, as the recruitment target of the older cohort was met).
* Participants may have been previously enrolled in the Compass Pilot but must have been discharged to routine screening. Women may also be in follow-up management for a previous abnormality or unsatisfactory cytology.

Exclusion Criteria:

* Previous total hysterectomy (uterus and cervix).
* The presence of symptoms or signs for which cervical cancer must be excluded.
* Currently undergoing treatment for cervical cancer.
* Currently enrolled in the Compass Pilot Study.

Ages: 25 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76181 (Actual)
Dates: Start 2015-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative CIN3+ (Cervical Intraepithelial Neoplasia Grade 3 or invasive cervical cancer) (ITT) | Expected 5 year follow-up
  The primary outcome will be cumulative CIN3+ at 5 years following a 5 year HPV exit testing round in both arms, in women randomised to the HPV arm vs. women randomised to the LBC arm, adjusted for censoring after CIN2+ treatment. For the primary outcome, intention to treat analysis will be performed with closed loop testing for non-inferiority and superiority if non-inferiority is declared. Assuming a total average CIN3+ rate in the LBC arm (across unvaccinated and vaccinated women) of 0.94%, and an absolute non-inferiority margin of 0.22%, the trial will have 78% power with 97.5% confidence to detect non-inferiority for the HPV arm, allowing for a 15% non-compliance rate.

SECONDARY OUTCOMES:
Cumulative CIN3+ in baseline screen-negative women (ITT) | Expected 5 year follow-up
  Cumulative CIN3+ in women presenting for routine screening randomised to the HPV arm who were HPV-negative at baseline, vs. CIN3+ in those randomised to the LBC arm and who were LBC-negative at baseline, adjusted for censoring after CIN2+ treatment and stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980). Intention to treat analysis will be performed with closed loop testing for non-inferiority and superiority if non-inferiority is declared.
Cumulative CIN3+ in baseline screen-negative women (per protocol) | Expected 5 year follow-up
  Cumulative CIN3+ in women presenting for routine screening randomised to the HPV arm who were HPV-negative at baseline, vs. CIN3+ in those randomised to the LBC arm and who were LBC-negative at baseline and at 2.5 years, adjusted for censoring after CIN2+ treatment and stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980). Per-protocol analysis will be performed in women screened and followed up within a defined tolerance period according to protocol recommendations.
Cumulative CIN2+ in baseline screen-negative women (ITT) | Expected 5 year follow-up
  Cumulative CIN2+ in women randomised to the HPV arm who were HPV-negative at baseline, vs. CIN2+ in women who were randomised to the LBC arm and were LBC-negative at baseline, adjusted for censoring after CIN2+ treatment and stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980).
Baseline CIN2+ and CIN3+ | Following recruitment
  Cross-sectional outcomes for CIN 2+ and CIN3+ detection in each arm, stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980).
CIN2+ in women randomised to HPV testing at baseline with other oncogenic HPV | Expected 12-24 month follow-up
  CIN2+ in women randomised to HPV testing at baseline who have other HPV (not 16/18), stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980).
CIN2+ and CIN3+ in women who have an abnormal test result at baseline | Expected 5 year follow-up
  CIN2+ and CIN3+ in women who have an abnormal test result at baseline, adjusted for censoring after CIN2+ treatment and stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980).
CIN2+ and CIN3+ in women who were in follow-management for a previous abnormality at baseline | Expected 5 year follow-up
  CIN2+ and CIN3+ in women who were in follow-management for a previous abnormality at baseline, adjusted for censoring after CIN2+ treatment and stratified by recruitment group (date of birth >=July 1st 1980 and <1st July 1980).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Canfell, BE, D.Phil., Principal Investigator — University of Sydney; Marion Saville, M.B., Ch.B, Principal Investigator — Australian Centre for the Prevention of Cervical Cancer
Locations (1):
- VCS Foundation, Carlton, Victoria, Australia

REFERENCES:
- [Background] Canfell K, Caruana M, Gebski V, Darlington-Brown J, Heley S, Brotherton J, Gertig D, Jennett CJ, Farnsworth A, Tan J, Wrede CD, Castle PE, Saville M. Cervical screening with primary HPV testing or cytology in a population of women in which those aged 33 years or younger had previously been offered HPV vaccination: Results of the Compass pilot randomised trial. PLoS Med. 2017 Sep 19;14(9):e1002388. doi: 10.1371/journal.pmed.1002388. eCollection 2017 Sep. PMID 28926579
- [Background] Velentzis LS, Egger S, Waller J, Jennett CJ, Brotherton JML, Smith MA, Bateson D, Rogers C, Pagotto A, Skinner R, Taylor N, Edge R, Saville M, Canfell K. Correlates of intention-to-attend and confirmed cervical screening attendance during the COVID-19 pandemic in Australia: Findings from Compass-PLUS, a prospective cohort study. Prev Med Rep. 2024 Aug 5;45:102849. doi: 10.1016/j.pmedr.2024.102849. eCollection 2024 Sep. PMID 39220611
- [Background] Canfell K, Saville M, Caruana M, Gebski V, Darlington-Brown J, Brotherton J, Heley S, Castle PE. Protocol for Compass: a randomised controlled trial of primary HPV testing versus cytology screening for cervical cancer in HPV-unvaccinated and vaccinated women aged 25-69 years living in Australia. BMJ Open. 2018 Jan 26;8(1):e016700. doi: 10.1136/bmjopen-2017-016700. PMID 29374658
- [Derived] Yuill S, Hall MT, Caruana M, Lui G, Velentzis LS, Smith MA, Wrede CD, Bateson D, Canfell K. Predicted impact of HPV vaccination and primary HPV screening on precancer treatment rates and adverse pregnancy outcomes in Australia 2010-2070: Modelling in a high income, high vaccination coverage country with HPV-based cervical screening. Vaccine. 2025 Apr 30;54:126986. doi: 10.1016/j.vaccine.2025.126986. Epub 2025 Mar 15. PMID 40090212
- [Derived] Joshy G, Thandrayen J, Koczwara B, Butow P, Laidsaar-Powell R, Rankin N, Canfell K, Stubbs J, Grogan P, Bailey L, Yazidjoglou A, Banks E. Disability, psychological distress and quality of life in relation to cancer diagnosis and cancer type: population-based Australian study of 22,505 cancer survivors and 244,000 people without cancer. BMC Med. 2020 Dec 1;18(1):372. doi: 10.1186/s12916-020-01830-4. PMID 33256726
- [Derived] Sarich P, Canfell K, Egger S, Banks E, Joshy G, Grogan P, Weber MF. Alcohol consumption, drinking patterns and cancer incidence in an Australian cohort of 226,162 participants aged 45 years and over. Br J Cancer. 2021 Jan;124(2):513-523. doi: 10.1038/s41416-020-01101-2. Epub 2020 Oct 11. PMID 33041337
- [Derived] Smith MA, Gertig D, Hall M, Simms K, Lew JB, Malloy M, Saville M, Canfell K. Transitioning from cytology-based screening to HPV-based screening at longer intervals: implications for resource use. BMC Health Serv Res. 2016 Apr 26;16:147. doi: 10.1186/s12913-016-1375-9. PMID 27112193
- See also: Guidelines for human papillomavirus DNA test requirements for primary cervical cancer screening in women 30 years and older — http://www.ncbi.nlm.nih.gov/pubmed/18973271
- See also: Compass Trial Website — http://www.compasstrial.org.au/